CLINICAL TRIAL: NCT02139930
Title: Project 2: Strategies for Reducing Nicotine Content in Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: U54 DA031659-P2; U54DA031659 (NIH)
Record Dates: First submitted 2014-05-12; First posted 2014-05-16 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Nicotine Dependence; Tobacco Smoking
Keywords: smoking; nicotine reduction
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking; Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Nicotine Control Group (Active Comparator): These subjects will smoke normal nicotine content Spectrum brand cigarettes for 20 weeks.
  Interventions: Behavioral: Normal Nicotine Control Group
- Immediate Nicotine Reduction Group (Experimental): This group will immediately be switched to smoking very low nicotine content (VLNC) Spectrum brand cigarettes. They will smoke these cigarettes for 20 weeks.
  Interventions: Behavioral: Immediate Nicotine Reduction Group
- Gradual Nicotine Reduction Group (Experimental): This group will smoke progressively lower nicotine content Spectrum brand cigarettes for a period of one month each until they end up smoking the same VLNC cigarettes as the immediate reduction group.
  Interventions: Behavioral: Gradual Nicotine Reduction Group

INTERVENTIONS:
Behavioral: Normal Nicotine Control Group — Participants will smoke experimental cigarettes for a period of 20-weeks.
  Arms: Normal Nicotine Control Group
Behavioral: Immediate Nicotine Reduction Group — Participants will smoke experimental cigarettes for a period of 20-weeks.
  Arms: Immediate Nicotine Reduction Group
Behavioral: Gradual Nicotine Reduction Group — Participants will smoke experimental cigarettes for a period of 20-weeks.
  Arms: Gradual Nicotine Reduction Group

SUMMARY:
The main goal of this project is to compare two different approaches to reducing levels of nicotine in cigarettes: an immediate reduction in nicotine content in cigarettes to non-addictive levels or a gradual reduction in nicotine content in cigarettes to non-addictive levels. These two approaches will then be contrasted to a group that continues to smoke cigarettes with nicotine content similar to conventional cigarettes.

DETAILED DESCRIPTION:
This project will be conducted to compare product use patterns and biomarkers of exposure between smokers who are assigned to a) gradual reduction in reduced nicotine content (RNC) cigarettes; b) immediate reduction to very low nicotine content (VLNC) cigarettes or c) normal nicotine content (NNC) cigarettes. The outcomes from this study will provide information on different approaches to reducing levels of nicotine in cigarettes and will determine the approach with the most optimal outcomes taking into account the balance between overall risk reduction (possibly maximized by abrupt switching) and compliance and acceptability (possibly maximized by gradual reduction of RNC cigarettes).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Daily smokers who smoke an average of at least five cigarettes per day for at least 1 year
3. Breath CO levels > 8 ppm (if ≤ 8 ppm, then NicAlert Strip level must indicate regular smoking)

Exclusion Criteria:

1. Planned quit date in the next 30 days
2. Currently seeking treatment for smoking cessation
3. Currently using nicotine replacement therapies or other pharmacotherapies as cessation aid (non-cessation intermittent use acceptable)
4. A quit attempt in the past 30 days resulting in greater than 3 days of abstinence
5. Using other tobacco products or e-cigarettes more than 9 days in the past 30 days
6. Significant unstable medical conditions (Any significant change in a serious medical condition occurring during the past 3 months including, cardiovascular disease, COPD, and cancer, as determined by the licensed medical professional at each site)
7. Unstable psychiatric conditions (Any significant change in psychiatric symptoms during the past 3 months as determined by the licensed medical professional at each site)
8. Schizophrenia and schizoaffective disorder
9. Psychiatric medication changes (e.g., new prescriptions, changes in dosages, or discontinuation of medications) in the past 3 months that was a result of negative changes in symptoms.
10. Positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, and PCP

    1. Marijuana will be tested for but will not be an exclusionary criterion.
    2. Participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded.
    3. Participants failing the toxicology screen will be allowed to re-screen once.
11. Blood alcohol level > 0.01

    a. Participants failing the blood alcohol screen will be allowed to re-screen once.
12. Binge drinking alcohol (more than 9 days in the past 30 days, 4/5 drinks per day (female/male))
13. Pregnant, trying to become pregnant or breastfeeding
14. Predominant use of 'roll your own cigarettes'
15. CO reading >80 ppm
16. Systolic BP greater than or equal to 160

    a. Participants failing for blood pressure will be allowed to re-screen once.
17. Diastolic BP greater than or equal to 100

    a. Participants failing for blood pressure will be allowed to re-screen once.
18. Systolic BP below 90 and symptomatic (dizziness, extreme fatigue, difficulty thinking, inability to stand or walk, feeling faint)

    a. Participants failing for blood pressure will be allowed to re-screen once.
19. Diastolic BP below 50 and symptomatic (dizziness, extreme fatigue, difficulty thinking, inability to stand or walk, feeling faint)

    a. Participants failing for blood pressure will be allowed to re-screen once.
20. Heart rate greater than or equal to 105 bpm

    a. Participants failing for heart rate will be allowed to re-screen once.
21. Heart rate lower than 45 bpm and symptomatic (dizziness, extreme fatigue, difficulty thinking, inability to stand or walk, feeling faint)

    a. Participants failing for heart rate will be allowed to re-screen once.
22. Indicating any suicidal ideation in the past month, suicide attempts in the past 5 years (if within past 5 to 10 years, requires physician approval), or score of >4 on the MINI suicide subscale
23. Household member enrolled in the study concurrently.
24. Inability to independently read and comprehend the consent form and other written study materials and measures because participants are required to complete parts of the protocol at home independently.
25. Participated in prior study that involved reduced nicotine content cigarettes.
26. Having participated in a research study during the past three months in a study that would impact baseline smoking or response to study products.
27. Currently taking the following anticonvulsant medications:

    1. Phenytoin [Brand Name: Dilantin]
    2. Carbamazepine [Brand Name: Tegretol, Carbatrol, Equetro, Epitol]
    3. Oxcarbazepine [Brand Name: Trileptal]
    4. Primidone [Brand Name: Mysoline]
    5. Phenobarbital
28. Currently taking the following medication:

    1. Bendamustine (Treanda)
    2. Clopidogrel (Plavix)
    3. Clozapine (Clozaril, FazaClo)
    4. Erlotinib (Tarceva)
    5. Flecainide (Tambocor)
    6. Fluvoxamine (Luvox)
    7. Irinotecan (Camptosar)
    8. Olanzapine (Zyprexa)
    9. Ropinirole (Requip)
    10. Tacrine (Cognex)
    11. Theophylline (Theo Dur, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
Toxicant exposure pattern: Expired air carbon monoxide | 20-week treatment period
  Between group comparison of expired air carbon monoxide (CO) values at week 20 using baseline CO values as a covariate.
Toxicant exposure pattern: Urinary phenanthrene tetroal (Phe) | 20-week treatment period
  Between group comparison of urinary phenanthrene tetroal values at week 20 using baseline values as a covariate.
Toxicant exposure pattern: Urinary mercapturic acids of acrolein | 20-week treatment period
  Between group comparison of urinary mercapturic acid level at week 20 using baseline values as a covariate.

SECONDARY OUTCOMES:
Nicotine exposure: Total nicotine equivalents (TNE) | End of treatment (Week 20)
  Between group comparison of urinary total nicotine equivalents at week 20 using baseline values as a covariate.
Other toxicant exposure: Tobacco specific nitrosamines-Total NNAL and NNN | End of treatment (Week 20)
  Between group comparison of urinary total NNAL and NNN levels at week 20 using baseline values as a covariate.
Effect biomarker: C-Reactive protein-high sensitivity as an inflammation biomarker | End of treatment (Week 20)
  Between group comparison of C-Reactive protein levels in serum at week 20 using baseline values as a covariate.
Measure of acceptability: Retention in study | End of treatment (Week 20)
  Between group comparison of early termination from the study.
Measure of acceptability: Non-compliance | End of treatment (Week 20)
  Between group comparison of use of non-study tobacco products.
Effect biomarker: 8-epi-PGF2α as a biomarker for oxidative stress | End of treatment (Week 20)
  Between group comparison of 8-epi-PGF2α at week 20 using baseline values as a covariate.
Effect biomarker: White blood cells count as inflammation biomarker | End of treatment (Week 20)
  Between group comparison of white blood cell count at week 20 using baseline values as a covariate.
Nicotine exposure: Urinary cotinine | End of treatment (Week 20)
  Between group comparison of urinary total nicotine equivalents at week 20 using baseline values as a covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donny, PhD, Principal Investigator — University of Pittsburgh
Locations (10):
- United States (10):
  - Mayo Clinic, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota Medical School Duluth, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - Oregon Research Institute, Eugene, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MDAnderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Hatsukami DK, Luo X, Jensen JA, al'Absi M, Allen SS, Carmella SG, Chen M, Cinciripini PM, Denlinger-Apte R, Drobes DJ, Koopmeiners JS, Lane T, Le CT, Leischow S, Luo K, McClernon FJ, Murphy SE, Paiano V, Robinson JD, Severson H, Sipe C, Strasser AA, Strayer LG, Tang MK, Vandrey R, Hecht SS, Benowitz NL, Donny EC. Effect of Immediate vs Gradual Reduction in Nicotine Content of Cigarettes on Biomarkers of Smoke Exposure: A Randomized Clinical Trial. JAMA. 2018 Sep 4;320(9):880-891. doi: 10.1001/jama.2018.11473. PMID 30193275